CLINICAL TRIAL: NCT05150886
Title: The Validity of the ROX Index in Predicting Intubation in Patients With Covid-19 Pneumonia
Status: Completed | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mesut DEMİRKÖSE, Specialist Physician, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2434
Record Dates: First submitted 2021-12-07; First posted 2021-12-09 (Actual); Last update posted 2022-04-15 (Actual); Status verified 2022-04

CONDITIONS: COVID-19 Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 68 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients at low risk of intubation: Patients with a ROX index of 4.88 and above measured at the 12th hour of hospitalization in the intensive care unit.
  Interventions: Diagnostic Test: rox index
- Patients at hihg risk of intubation: Patients with a ROX index of less than 4.88, measured at the 12th hour of admission to the intensive care unit.
  Interventions: Diagnostic Test: rox index

INTERVENTIONS:
Diagnostic Test: rox index — After HFNC during reassessment, the ROX Index can help suggest which patients will fail HFNC and need to progress to intubation for further ventilatory support.

SUMMARY:
BACKGROUND: ROX index (SpO2 / FiO2) / respiratory rate, which is the ratio of peripheral oxygen saturation (SpO2) and inspired oxygen fraction (FiO2) divided by respiratory rate, to predict failure of HFNO therapy and intubation in patients with a rapid, easy-to-use, rapidly administered pneumonia. index used not to delay. This is a rating. HFNO reduces the need for endotracheal intubation in patients with acute hypoxic respiratory failure due to pneumonia. It has been suggested that HFNO may reduce the need for invasive mechanical ventilation compared to conventional oxygen therapy. Recently, experience has been reported that HFNO therapy also reduces the need for endotracheal intubation in patients with COVID-19 pneumonia. However, there are studies showing that insisting on HFNO and delaying intubation increase mortality in patients with acute respiratory distress syndrome (ARDS) and acute respiratory failure. In this study; We aimed to investigate the validity of the ROX index in predicting HFNO failure in patients with COVID-19 pneumonia admitted to the intensive care unit.

DETAILED DESCRIPTION:
BACKGROUND: ROX index (SpO2 / FiO2) / respiratory rate, which is the ratio of peripheral oxygen saturation (SpO2) and inspired oxygen fraction (FiO2) divided by respiratory rate, to predict failure of HFNO therapy and intubation in patients with a rapid, easy-to-use, rapidly administered pneumonia. index used not to delay. This is a rating. HFNO reduces the need for endotracheal intubation in patients with acute hypoxic respiratory failure due to pneumonia. It has been suggested that HFNO may reduce the need for invasive mechanical ventilation compared to conventional oxygen therapy. Recently, experience has been reported that HFNO therapy also reduces the need for endotracheal intubation in patients with COVID-19 pneumonia. However, there are studies showing that insisting on HFNO and delaying intubation increase mortality in patients with acute respiratory distress syndrome (ARDS) and acute respiratory failure. In this study; We aimed to investigate the validity of the ROX index in predicting HFNO failure in patients with COVID-19 pneumonia admitted to the intensive care unit.

MATERIAL - METHOD: The population of the research consists of patients who will be hospitalized in the COVID-19 intensive care unit of Health Sciences University Ankara Atatürk Chest Diseases and Thoracic Surgery Training and Research Hospital for 3 months. According to a study conducted in Italy, 87% of COVID-19 patients hospitalized in intensive care go to intubation (6). Adult patients (≥18 years old) with acute respiratory failure due to COVID-19 pneumonia, positive PCR on nasopharyngeal swab, and HFNO when admitted to the intensive care unit will be included in this study. Patients under the age of 18 who received non-invasive or invasive mechanical ventilation therapy before HFNO will not be included in the study. Patients with chronic lung disease will be excluded from the study. RT-PCR tests will be performed with serial samples for detection of viral RNA. Demographic, clinical, treatment and laboratory data of the patients will be recorded. ROX score, APACHE 2 scores, Pneumonia Severity Index (PSI) score, CURB-65 and SOFA score will be calculated and recorded. In addition, the day of hospitalization in the intensive care unit, intensive care and hospital mortality, intubation time, invasive mechanical ventilation day, time of exit from the intensive care unit and discharge from the hospital will be recorded.

ORGANİZATİON AND ANALYSİS OF RESEARCH DATA The sample number of the study was calculated with the OpenEpi online computer program. The number of samples calculated with α= 0.05, d=5 and 87% frequency in the 95% confidence interval is 122. SPSS 23.0 statistical package program will be used for statistical analysis of research data. As a statistical analysis, in the descriptive findings section, categorical variables will be presented as numbers and percentages, and continuous variables will be presented as mean±standard deviation (min-max) for data showing normal distribution and median (IQR; 25-75). For categorical variables for non-normally distributed data, whether there is a frequency difference between groups will be compared using appropriate chi-square tests. Continuous variables will be compared with the normal distribution using Student's t test or Mann-Whitney U test. ROC analysis will be performed to determine whether the ROX index has a good cut-off value in making the intubation decision of COVID-19 patients. Statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years of age) with acute respiratory failure due to COVID-19 pneumonia, PCR positive in the nasopharyngeal swab, and HFNO on admission to the intensive care unit will be included in this study.

Exclusion Criteria:

* Patients under the age of 18 who received non-invasive or invasive mechanical ventilation therapy before HFNO will not be included in the study. Patients with chronic lung disease will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the intensive care unit.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-08 (Actual)

PRIMARY OUTCOMES:
intubation | 3 month
  We aimed to investigate the validity of the ROX index in predicting HFNO failure in patients with COVID-19 pneumonia admitted to the intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: MESUT DEMİRKÖSE, Principal Investigator — university
Locations (1):
- MESUT, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The Validity of the ROX Index in Predicting Intubation in Patients with Covid-19 Pneumonia
Supporting Information: Study Protocol
Time Frame: It will be available for 4 months as of February 1, 2022
Access Criteria: The datasets generated during and/or analysed during the current study will be stored in a non-publically available repository.